CLINICAL TRIAL: NCT00967512
Title: Aezea (Cenersen) in Combination With Chemotherapy for Treatment of Acute Myelogenous Leukemia Subjects ≥55 Years of Age With No Response to Single Frontline Induction Course in a Randomized Double-Blind Placebo-Controlled Multi-Center Study
Brief Title: Aezea® (Cenersen) and Chemotherapy for AML Subjects ≥ 55 Years of Age With No Response to Frontline Induction Course
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Was Terminated due to lack of Funding.
Sponsor: Eleos, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ELP1020; 2008-002160-34 (EudraCT Number)
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Oligonucleotides, Antisense; Tumor Suppressor Protein p53; idarubicin; cytarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — cenersen; Sodium Chloride; Idarubicin; Cytarabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- cenersen, idarubicin, cytarabine (Experimental): cenersen, idarubicin, cytarabine
  Interventions: Drug: cenersen; Drug: idarubicin, cytarabine
- placebo, idarubicin, cytarabine (Placebo Comparator): placebo, idarubicin, cytarabine
  Interventions: Drug: placebo; Drug: idarubicin, cytarabine

INTERVENTIONS:
Drug: cenersen — solution for injection, intravenous infusion, 0.1 mg/kg/h x 24h x 4 days, and 0.4 mg/kg/h x 3h x 4 days
  Other Names: Aezea®; cenersen sodium; EL625
  Arms: cenersen, idarubicin, cytarabine
Drug: placebo — solution for injection, intravenous infusion, 0.1 mg/kg/h x 24h x 4 days, and 0.4 mg/kg/h x 3h x 4 days
  Other Names: saline
  Arms: placebo, idarubicin, cytarabine
Drug: idarubicin, cytarabine — idarubicin, cytarabine
  Other Names: idamycin; Ara-C

SUMMARY:
The purpose of this study is to assess whether treatment with cenersen in combination with 4 cycles of high and low-dose chemotherapy (idarubicin and cytarabine) improves the complete response rate in acute myelogenous leukemia (AML) patients ≥ 55 years of age who did not show a response (CR, CRi, or PR) to a single aggressive frontline induction course.

DETAILED DESCRIPTION:
Cenersen is a phosphorothioate antisense oligonucleotide of sequence 5'-CCCTG5-CTCCC10-CCCTG15-GCTCC20-3'. For AML, cenersen is specific for blocking p53 expression in the stem cells. When AML stem cells are dividing, cenersen sensitizes them to even low-level DNA damage of the type caused by idarubicin, etoposide and possibly ara-C.

Because AML stem cells are not all dividing at any given time, this protocol is designed to treat patients with a total of four cycles of cenersen plus chemotherapy within a two to three month period. For a limited period of time, proliferating non-stem cells can be expected to maintain or even expand the tumor while the stem cells are being depleted. If the proliferating non-stem cells are not resupplied by the stem cells, they will all become end stage blasts after a few divisions and undergo elimination.

ELIGIBILITY:
Inclusion Criteria:

* In response to their first course of frontline treatment, patients who did not achieve a response (CR, CRi, or PR) and have ≥ 15% bone marrow blasts in a BM specimen between day 14 - 42 from the initiation of a single frontline course. If within that timeframe the BM is hypoplastic, the BM assessment can be repeated within a subsequent two-week period and the patient entered into the study if there is ≥ 15% blasts in the bone marrow.
* ≥ 55 years old
* Have an understanding of the importance of not taking paracetamol (acetaminophen) or high dose antioxidants from 1 day before through 1 day after treatment during any given course
* Have a life expectancy of more than 4 weeks following initiation of treatment
* Secondary AML is allowed as are antecedent hematologic disorders
* Zubrod performance status ≤ 2
* Have recovered from acute toxicities of prior chemotherapy (≤ Grade 2)
* Have signed an informed consent
* Total bilirubin ≤ 1.5 x upper normal limit (UNL) and Alanine Amino Transferase [ALT (Serum Glutamic-pyruvic Transaminase (SGPT))] ≤ 2.5 x UNL
* Creatinine ≤ 1.5 x UNL
* Serum magnesium should be within the normal range (Mg replacement being acceptable)
* Left Ventricular Ejection Fraction (LVEF) of >50% as determined by multiple-gated acquisition scan (MUGA) or Echocardiogram (ECHO)
* Ability to receive all courses of therapy, as outlined in the treatment schedules at the investigative site
* Willingness to comply with scheduled follow-up as required by the protocol
* Use of adequate contraceptive techniques if premenopausal and sexually active; examples include implantable, injectable or oral contraceptives, intrauterine devices (IUD), sterilization, or sexual abstinence
* If premenopausal, have negative pregnancy tests at screening

Exclusion Criteria:

* Presence of any pneumonia regardless of severity or other life-threatening illness including, but not limited to, ongoing infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, high blood pressure, history of labile hypertension, history of poor compliance with an antihypertensive regimen, myocardial infarction less than or equal to 6 months prior to registration, diabetes, or extensive and symptomatic interstitial fibrosis of lung, chronic liver disease or psychiatric illness/social situations that limits compliance with study requirements
* Acute promyelocytic leukemia (APL [FAB classification M3])
* Requirement for transplant before Course 2 is complete
* Concurrent use of other experimental agents (i.e., drugs not approved for clinical indications) or having received other investigational agents within the 30 days prior to the start of Course 1
* Pregnancy (includes a positive pregnancy test at the screening visit) or lactation
* Known HIV infection
* Active hepatitis B or C or other active liver disease
* Presence of dyspnea at rest or with minimal exertion after correction for anemia
* Known or suspected hypersensitivity or allergy to idarubicin or ara-C
* Occurrence of major surgery within two weeks of the start of Course 1
* Chemotherapy within two weeks prior to initiation of therapy under this protocol, or hydroxyurea within 7 days
* Patients who, with appropriate explanation, are not prepared to exclude the use of paracetamol (acetaminophen) or paracetamol-containing medications from 1 day before through 1 day after treatment during any course
* Patients who are not prepared to commit to the exclusion of high dose antioxidants from 1 day before through 1 day after treatment during any given course
* Medical or psychiatric conditions that compromise the ability to give informed consent, to comply with the protocol or to complete the study
* Inability, in the opinion of the principal investigator or clinical staff, to comply with protocol requirements for the duration of the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Complete Remission Rate | within day 28-42 of Course 1, and within day 28-42 of Course 2

SECONDARY OUTCOMES:
Overall Survival | 2 years
Safety Profile | up to 2 years
Complete Remission + Complete Remission with Incomplete Blood Count Recovery Rate | within day 28-42 of Course 1, and within day 28-42 of Course 2
Morphologic Leukemia-Free State Rate | within day 28-42 of Course 1, and within day 28-42 of Course 2
Partial Remission Rate | within day 28-42 of Course 1, and within day 28-42 of Course 2
Remission Duration | 2 years
Early deaths measured as deaths at 30, 60 and 90 days of the start of treatment | 30, 90, and 90 days from start of treatment
Time to Neutrophil and Platelet Recovery | within day 28-42 of Course 1, and within day 28-42 of Course 2
Death in Complete Remission | 2 years
Zubrod Score | during Frontline Assessment (screening); Course 1: on days 6, 15, 18, and within day 28-42; Course 2: on days 1, 7, 15, 18, and within day 28-42; Course 3: on days 1 and 6; and Course 4: on days 1 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Larry J Smith, PhD, Study Chair — Eleos, Inc.